CLINICAL TRIAL: NCT05375227
Title: Assessment of a Sonic Toothbrush on the Abrasion of the Gingival Tissue
Acronym: ASTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Philips France Commercial (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2020-A02614-35
Record Dates: First submitted 2021-10-26; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Gingival Abrasion

STUDY DESIGN:
Intervention Model Description: A randomized, monocentric, examiner-blind, two-arm, parallel, controlled clinical research study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electric Toothbrush (Experimental): Electric toothbrush + manufacturer's instructions + professional recommendations + sodium monofluorophosphate (1450 ppm F) toothpaste (elmex® SENSITIVE PROFESSIONAL)
  Interventions: Other: Teeth brushing
- Manual toothbrush (Active Comparator): Manual toothbrush + manufacturer's instructions + professional recommendations + sodium monofluorophosphate (1450 ppm F) toothpaste (elmex® SENSITIVE PROFESSIONAL)
  Interventions: Other: Teeth brushing

INTERVENTIONS:
Other: Teeth brushing — The participants will be invites to brush their teeth twice a day for 3 months using either an electric toothbrush or a mannual toothbrush and low abrasivity toothpaste

SUMMARY:
This is a randomized, monocentric, examiner-blind, two-arm, parallel, controlled clinical research study. It aims to assess gingival abrasion by the comparison of pre- to- post-brushing after a single brushing and after 12 weeks of daily home brushing using a macro-relief scoring based on photographs of the gingiva. The study also aims to assess plaque removal, gingival inflammation, gingival recession and gingival color after 12 weeks. To enter the study, adult male and female subjects attending the service of odontology at Rothschild hospital (Paris, France) will refrain from all oral hygiene procedures for 24 hours. Subjects will have the study procedure explained to them both orally and by written instructions. Eligible patients will give their written consent to participate before being included into the study. Following a baseline clinical examination for collection of the following periodontal parameters: plaque control record (PCR), bleeding on probing (BOP), gingival recession (REC), and probing pocket depths (PD), the subjects will be randomized into two balanced groups, test group assigned to the Sonicare ProtectiveClean® HX6848/92 with C2 Optimal Plaque Defense head HX9022/10 (electric toothbrush) and control group assigned to the Pierre Fabre Inava 20/100, a reference manual toothbrush. Subjects will be instructed to brush their teeth for one minute under supervision with their assigned toothbrush and a sodium monofluorophosphate (1450 ppm F) toothpaste (elmex® SENSITIVE PROFESSIONAL) with a low level of abrasion to minimize bias due to toothpaste abrasivity. After brushing, they will again be evaluated for primary and secondary outcomes (post-brushing). Subjects will be dismissed from the study site with their assigned toothbrush and toothpaste, and instructed to brush twice daily at home for the next 12 weeks. The subjects will be instructed to brush for two minutes during each tooth brushing. The subjects will report to the study site after 12 weeks of product use, at which time they will be re-evaluated for gingival abrasion, as well as for plaque removal, gingival inflammation, gingival recession and gingival color. Data (photographs and clinical measurements) will be collected, i.e. primary and secondary variables of each patient, by blinded examiners.

ELIGIBILITY:
Inclusion Criteria:

1. Dentate males and females must be at least 18 years and not more than 75 years of age
2. Patient able to understand and sign the informed consent prior to starting the study
3. Patient with a minimum of 3 teeth in each of the 4 quadrants and no/or pockets >4 mm
4. Ability and willingness to comply with all study requirements.

Exclusion Criteria:

1. Pregnancy
2. Patient with cervical restorations
3. Current smoker
4. Patient with orthodontic banding
5. Patient with oral lesions or periodontal diseases
6. Patient who has been deprived of his/her freedom by administrative or legal decision or who is under trusteeship/guardianship
7. Patient already using an electric toothbrush
8. Patient with conditions or circumstances, which may prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance, or unreliability;
9. Patient with non-plaque induced gingival diseases or localized gingival ulceration
10. Thin gingival phenotype
11. Patients with cardiac pacemakers to prevent any interference between the power toothbrush and the implantable cardiac device.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the gingival abrasion (GA): Macro-relief scoring | 90 days
  A first method for the evaluation of gingival abrasion (GA) will consist in a method of macro-relief scoring of gingival tissue as described previously by Perin et al. with skin tissue. This evaluation consists of acquiring macroscopic views of each investigated surface and then classifying them by observers according to a reference groups of defined abrasion intensity. This evaluation scoring, using photo grading technique, allow delayed and blinded scoring, independent of whole-subject appearance, thus decreasing subjectivity (Perin et al., 2000).
  Five items are evaluted for each picture : erythema, inflammation, bleeding, recession and erosion of the gingiva. All items are scored from 0 to 3, 3 representing the most significant impairment.

SECONDARY OUTCOMES:
Comparison of gingival color; | 90 days
  Comparison of gingival color between baseline and time point using photographs. The technique consists of acquiring macroscopic photographs of each gingival quadrant, including an internal colored reference chart in the vicinity of the photographed gingival tissue, at each time point. Next, using an image analysis software, each photograph will be calorimetrically reconverted to be recalibrated following the colored reference chart. Then, the coloring intensity in each zone of interest [marginal (cervical free gingiva, CFG), interdental (papillary free gingiva, PFG) and mid-gingival (attached gingiva, AG)] around each tooth in each quadrant, will be extracted by observers in a double-blind manner using the color picker tool.
  This method has already been applied to describe the intensity of skin coloring (red /green/blue component) as well as luminosity, the brightness and transparency (Musnier et al., 2004) and will be applied to each subject's gingival tissue.
Presence of plaque -Plaque index, PI | 90 days
  Plaque index (PI) described by Silness & Löe (Silness and Löe, 1964) uses 0 to 4 classes to assess the presence of plaque or not on six sites (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual, and disto-lingual) on all teeth, according to the following criteria: 0: absence of plaque; 1: non visible plaque but detectable with a probe; 2: visible plaque not detectable in the interproximal areas; 3: visible plaque in interdental spaces also.
Presence of inflammation BOP | 90 days
  Gingival inflammation (GI) will be assessed as bleeding on marginal probing (BOP) using the index as described by Ainamo & Bay (Ainamo and Bay, 1975). GI uses a 0 to 3 scale to measure the presence of inflammation or not on six sites (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual, and disto-lingual) on all teeth, according to the following criteria: 0: absence of inflammation; 1: visible inflammation and no bleeding; 2: visible inflammation and bleeding on probing; 3: obvious inflammation and spontaneous bleeding.
  BOP is considered as dichotomous variable. BOP uses 0 and 1 scale. 0: no bleeding on probing; 1: bleeding on probing including 4 sites per tooth. The percentage of bleeding will be calculated as following: number of sites with bleeding / number of sites assessed X 100.
Presence and/or amount of gingival recession (REC) | 90 days
  Gingival margin recession will be measured from the cemento-enamel junction to the marginal position of the gingiva with PCP-UNC 15 (Hu-Friedy® Chicago, IL, USA) probe. The measurements will be assessed at the middle of the buccal gingival recession.
Probing pocket depth (PD) | 90 days
  PD will be measured before the test/control treatment by one and the same examiner by using the PCP-UNC 15 (Hu-Friedy® Chicago, IL, USA) probe throughout the study. The probing depth will be assessed at the buccal aspects of teeth 16,14,13,11. All measurements will be adjusted to the nearest 1.0 mm.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe BOUCHARD, Pr Dr, Principal Investigator — Rothschild Hospital
Locations (1):
- Rothschild Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/27/NCT05375227/Prot_000.pdf